CLINICAL TRIAL: NCT06404229
Title: Novel Use of Bedside Arm Ergometry CardioPulmonary Exercise Tests for the Risk Stratification of Patients With Chronic Limb-threatening Ischaemia: A Feasibility Trial
Brief Title: Use of CPETarm for Risk Stratification of Patients With CLTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jonathan Ghosh, Honorary Reader Cardiovascular Sciences, Consultant and Clinical Director, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 329960
Record Dates: First submitted 2024-03-12; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Chronic Limb-Threatening Ischemia; Surgery-Complications
Keywords: CardioPulmonary Exercise Testing; Risk Stratification
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CardioPulmonary Exercise Testing (Experimental): All patients included in the study will perform CardioPulmonary Exercise Testing prior to surgery
  Interventions: Diagnostic Test: CardioPulmonary Exercise Testing

INTERVENTIONS:
Diagnostic Test: CardioPulmonary Exercise Testing — CardioPulmonary Exercise Testing using an arm ergometer prior to surgery

SUMMARY:
This is a prospective cohort study of patients undergoing surgery for chronic limb threatening ischaemia. Prior to surgery, patients will undergo CardioPulmonary Exercise testing (CPET) using an arm ergometer. Feasibility outcome measures will be recorded at testing and participants will be followed up for a period of up to 5 years to obtain clinical outcome measures.

DETAILED DESCRIPTION:
Chronic limb-threatening ischaemia (CLTI) is the most severe clinical manifestation of peripheral arterial disease, defined by the presence of pain at rest and/or tissue loss affecting the legs. It is a major cause of chronic pain, amputation and death. CLTI is a growing global healthcare problem attributable to the ageing population and increase of risk factors such such as diabetes.

Prevalence of high blood pressure, heart disease and diabetes is high amongst this cohort of patients and so it is unsurprising that surgery is associated with an alarmingly high risk of illness, complications and even death when compared to other types of surgery. As nearly half of the patients present as an emergency, assessment and optimisation of health prior to surgery is challenging.

The aims of the assessment prior to surgery includes optimising any current health problems, understanding what care may be required after surgery, allowing the patient to be fully informed of the risks and considering non surgical options where appropriate. Inadequate risk stratification can lead to delays in theatre, increased length of hospital stay and unnecessary loss of limb and/or life.

Currently there is no established method to risk stratify CLTI patients presenting as an emergency. CardioPulmonary Exercise Testing (CPET) is an exercise test useful in identification of a number of heart and lung conditions. The test is established for risk-stratification in other populations but its method of using a bicycle is not suitable for CLTI patients, nor has it previously been used in the emergency setting. This study will assess whether CPET using arm exercise instead of the traditional bicycle is a feasible test that can be performed at the bedside within 48 hours of intention to treat, required to make it a practical test in the assessment of emergency patients.

Hypothesis:

1. Cardiopulmonary exercise testing using an arm ergometer (CPETarm) is a feasible, acceptable and safe tool to use at the 'bedside' in patients undergoing emergency surgery for chronic limb threatening ischaemia (CLTI).
2. Values obtained from CPETarm and/or hand grip strength can be used to predict post operative outcomes including major adverse cardiovascular events and mortality for this group of patients.

Recruitment:

The study will enrol 120 consecutive, eligible and consenting patients admitted with with CLTI to the Manchester Vascular Centre at Manchester University National Health Service Foundation Trust. Patients scheduled to undergo non elective surgical or endovascular treatment of their chronic limb threatening ischaemia will be screened for inclusion. Decision for surgery/management will be recommended by their Consultant Vascular Surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written informed consent
* Diagnosis of chronic limb threatening ischaemia, undergoing one of the following procedures: Infra inguinal bypass, Extra anatomical bypass, Common femoral endarterectomy, Endovascular treatment, Primary amputation

Exclusion Criteria:

* Patients with active medical conditions deemed an absolute contraindication for undertaking CPET
* Ongoing evaluation for coronary artery disease (e.g awaiting stress test or cardiac catheterisation or requiring the up titration of anti anginal medications)
* Active arrthymic requiring the initiation or up titration of an anti arrthymic medication
* Active congestive cardiac failure requiring the initiation or up titration of diuretic therapy.
* Severe cardiac valvular stenosis
* Physical disability precluding ability to perform CPETarm
* Psychiatric disorder or dementia precluding them from consenting for research and/or undertaking testing and/or follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-28 (Estimated); Primary Completion 2025-05-28 (Estimated); Study Completion 2030-04-28 (Estimated)

PRIMARY OUTCOMES:
Acceptability of bedside CPET | At time of CPET testing (1 day)
  The percentage of recruited participants actually performing CPET compared to the number of patients consenting.
  (A) identifying reasons, and their number, as to why participants did not undertake CPET, and (B) identifying reasons, and their number, for clinician-led termination of CPET
Recruitment rate (uptake of bedside CPET) | At time of CPET testing (1 day)
  The percentage of eligible patients who gave informed consent to participate in the study
Practicality of bedside CPET | At time of CPET testing (1 day)
  Recorded as three variables
  1. Time between decision for surgical intervention and CPET testing
  2. Location of testing
  3. Duration of testing (inclusive of set up, patient instructions, completion of test and recovery)
Patient reported outcome measures | 30 days
  Established by identifying participant opinions on satisfaction with, and suitability of, CPET for future use.
  Assessed in a qualitative manner using a semi structured interview with 8 pre determined questions and quantitatively using a 5 point Likert scale for 12 statements, whereby 1='strongly disagree' and 5='strongly agree'.
Adverse or unexpected events report | At time of CPET testing (1 day)
  Defined as participants experiencing serious adverse events during or after the test.
  Defined adverse events for CPET as: 1) death during the stress test, 2) external defibrillation or implantable cardioverter-defibrillator discharge, 3) sustained ventricular tachycardia (wide complex tachycardia lasting longer than 30 seconds), 4) myocardial infarction, 5) syncope, 6) administration of advanced cardiac life support medications, 7) referral for direct hospital admission, or 8) referral to emergency department

SECONDARY OUTCOMES:
Peri-operative complications | Recorded at 30 days
  Defined as defined as any complication that occurred during surgery or within 30 days of surgery. Graded using the Clavien-Dindo classification.
All cause mortality | Recorded at 30 days, 90 days, 1 year, 3 years and 5 years
  Defined as death from any cause during the study
Amputation-free survival | Recorded at 30 days, 90 days, 1 year, 3 years and 5 years
  Freedom of death and major limb amputation during the study
Level of care post-surgery | Recorded at 30 days
  Categorised as according to the ward the patient is cared for in the immediate post operative period.
  * Level 0 (postoperative recovery on a surgical ward
  * Level 1 (postoperative recovery on a surgical ward with access to a critical care outreach team)
  * Level 2 (high dependency unit, post anaesthesia care unit)
  * Level 3 (intensive care unit)
Higher level of care length of stay | Recorded at 30 days
  Recorded as the length of stay on a ward categorised as level 2 or 3.
Length of hospital stay | Recorded at 30 days
  Defined as number of days spent in index hospital from date of operation.
Discharge destination | Recorded at 30 days
  Recorded as place of discharge from hospital. Discharge destination, dichotomized as home or non-home. Non-home discharge was defined as discharge to a skilled care facility (e.g., a transitional care unit, subacute hospital, or skilled nursing home), unskilled care (e.g., nursing home or assisted facility, only if this was not the patient's preoperative location), separate acute care, rehabilitation, or a multi-level senior community)
Rate of re-intervention | Recorded at 30 day and 90 days
  Primary patency: Freedom from occlusion of bypass-graft or endovascular treated arterial segment and freedom of restenosis that need intervention in bypass-graft or endovascular treated arterial segment.
  Secondary patency: Freedom from occlusion of bypass-graft or endovascular treated arterial segment. Treated for restenosis in bypass-graft or endovascular treated arterial segment.
Hospital readmission rate | Recorded at 30 and 90 days.
  Defined as a readmission after discharge from the index hospital stay and within 90 days of the primary surgical procedure
Health related quality of life | Recorded at 30 and 90 days
  Health related quality of life measured by The Vascular Quality of Life Questionnaire 25 (VASCUQOL25). VascuQol consists of 25 items, subdivided into five domains. Each question has a seven-point response scale. The responses are averaged to give an overall and a domain score ranging from one (worst Health Related Quality of Life, HRQoL) to seven (best HRQoL).
Major adverse cardiovascular events | Recorded at 30 and 90 days
  Defined as non fatal myocardial infarction, non fatal stroke, cardiovascular death, coronary intervention or unstable angina requiring hospitalisation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] [1] Conte MS, Bradbury AW, Kolh P, et al. GVG Writing Group for the Joint Guidelines of the Society for Vascular Surgery (SVS), European Society for Vascular Surgery (ESVS), and World Federation of Vascular Societies (WFVS). Global Vascular Guidelines on the Management of Chronic Limb-Threatening Ischemia. Eur J Vasc Endovasc Surg. Eur J Vasc Endovasc Surg, 2019. 58: p. 1-109.
- [Background] [2] Waton S, Johal A, Li Q, et al. National Vascular Registry: 2023 State of the Nation Report. London: The Royal College of Surgeons of England, November 2023.